CLINICAL TRIAL: NCT05093790
Title: A Phase 2a Single Dose Study to Evaluate the Effect of BMS-986141 Added on to Aspirin or Ticagrelor or the Combination, on Thrombus Formation in an Ex Vivo Thrombosis Chamber Model in Patients With Stable Coronary Artery Disease and Healthy Participants
Brief Title: A Study to Evaluate BMS-986141 Added on to Aspirin or Ticagrelor or the Combination, on Thrombus Formation in a Thrombosis Chamber Model in Participants With Stable Coronary Artery Disease and Healthy Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV006-037; 2020-005209-18 (EudraCT Number)
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Healthy Participants
Keywords: Thrombosis; Coronary Artery Disease; Healthy Participants; Aspirin; Ticagrelor; Brilinta; BMS-986141
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis | interventions — Ticagrelor; BMS-986141; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment Arm 1: Ticagrelor + BMS-986141 (Experimental)
  Interventions: Drug: Ticagrelor; Drug: BMS-986141
- Treatment Arm 2: Aspirin + BMS-986141 (Experimental)
  Interventions: Drug: BMS-986141; Drug: Aspirin
- Treatment Arm 3: Ticagrelor + Aspirin + BMS-986141 (Experimental)
  Interventions: Drug: Ticagrelor; Drug: BMS-986141; Drug: Aspirin
- Treatment Arm 4: BMS-986141 (Experimental)
  Interventions: Drug: BMS-986141

INTERVENTIONS:
Drug: Ticagrelor — Specified dose on specified days
  Other Names: Brilinta
  Arms: Treatment Arm 1: Ticagrelor + BMS-986141; Treatment Arm 3: Ticagrelor + Aspirin + BMS-986141
Drug: BMS-986141 — Specified dose on specified days
Drug: Aspirin — Specified dose on specified days
  Other Names: Acetylsalicylic acid (ASA)
  Arms: Treatment Arm 2: Aspirin + BMS-986141; Treatment Arm 3: Ticagrelor + Aspirin + BMS-986141

SUMMARY:
The purpose of this study is to assess the effectiveness, safety and tolerability of BMS-986141 added on to aspirin or ticagrelor or the combination on thrombus formation in both healthy participants and participants with stable coronary artery disease.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit: www.BMSStudyConnect.com

Inclusion Criteria:

* Male or female between 18 to 75 years of age, inclusive, and body mass index (weight kg/m2) between 18 and 35 kg/m2 (inclusive), and body weight 50 kg and 120 kg (inclusive)
* Judged to be generally in good health based on medical history, physical examination, ECGs, vital signs and laboratory tests
* Signed an informed consent document indicating they understand the purpose of and procedures required for the experiment and are willing to participate in the experiment
* Willing/able to adhere to the visit schedule
* For treatment arms groups with stable CAD participants (not for healthy volunteers without CAD) one or more of: Prior angiographically proven CAD (>50% stenosis of proximal coronary artery), prior coronary revascularization (PCI or CABG), prior myocardial infarction (MI)

Exclusion Criteria:

* Participants who meet any of the following criteria will be excluded from participating in the experiment: Allergies or intolerance of aspirin, ticagrelor and BMS-986141, requirement for dual antiplatelet therapy, requirement for anticoagulant therapy
* Acute Coronary syndrome or coronary revascularization within 3 months
* Coagulation disorders (including any abnormal bleeding or blood dyscrasias), anemia, renal or hepatic insufficiency or any others illness that the investigator considers should exclude the participants/patients of that could interfere with the interpretation to the results
* Acute illness, including a common cold, within 7 days prior to visit or other significant acute or chronic medical illness
* Major or traumatic surgery within 12 weeks of screening
* History of, a reason to believe that, a blood donor subject has a history of drug or alcohol abuse within the past 5 years or has not abstained from alcohol for at least 24 hours prior to visit
* Positive serum or urine pregnancy test
* Not anatomically suitable for or unwilling to undergo venipunctures
* Participation in a study of an investigational medicinal product within the last 4 weeks
* Any condition that, in the opinion of the investigator, would compromise the wellbeing of the blood donor subject or the experiment or prevent the blood donor subject from meeting or performing experiment requirements

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Nash J, Meah MN, Whittington B, Debono S, Raftis J, Miller MR, Sorbie A, Mills NL, Nespoux J, Bruce L, Duffin R, Dhaun N, Brittan M, Chao L, Merali S, Kim M, Wang Z, Zhang Y, Jin S, Wang B, Kozinn M, Newby DE. PAR4 Antagonism in Patients With Coronary Artery Disease Receiving Antiplatelet Therapies. Arterioscler Thromb Vasc Biol. 2024 Apr;44(4):987-996. doi: 10.1161/ATVBAHA.123.320448. Epub 2024 Feb 15. PMID 38357820
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 58 participants received study treatment
Groups:
- Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141: Single oral dose of 90 mg ticagrelor alone, followed by a single oral dose of 4 mg BMS-986141 approximately 2 hours later (Day 1). A second dose of ticagrelor will be taken approximately 12 hours after the first dose. Twice daily dosing of ticagrelor will be continued on Day 2.
- Arm 2: 75 mg Aspirin + 4 mg BMS-986141: Single oral dose of 75 mg aspirin alone, followed by a single oral dose of 4 mg BMS-986141 approximately 2 hours later (Day 1). Daily dosing of aspirin will continue on Day 2.
- Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141: Single oral dose of 90 mg ticagrelor + 75 mg aspirin, followed by a single oral dose of 4 mg BMS-986141 approximately 2 hours later (Day 1). A second dose of ticagrelor will be taken approximately 12 hours after the first dose. Ticagrelor + aspirin dosing will continue on Day 2.
- Arm 4: Heathy Participants: Heathy Participants received a single dose of 4 mg BMS-986141 on Day 1.
Period: Overall Study
Arm/Group | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 | Arm 4: Heathy Participants
Started | 16 | 15 | 16 | 11
Completed | 15 | 15 | 15 | 11
Not Completed | 1 | 0 | 1 | 0
Not completed — Failure to meet continuation criteria | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 | Arm 4: Heathy Participants | Total
Number analyzed (Participants) | 16 | 15 | 16 | 11 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (5.4) | 66.3 (7.6) | 62.3 (6.1) | 31.0 (11.9) | 58.3 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 0 | 3 | 10
  Male | 12 | 12 | 16 | 8 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 16 | 15 | 16 | 11 | 58
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Thrombus Area
Description: The change from baseline in thrombus area post-treatment with BMS-986141 versus pretreatment. Baseline is defined as the last non-missing result (including repeated and unscheduled assessments) with a collection date-time less than the datetime of study medication.
Time Frame: Baseline, Day 1 hour 2, Day 2 hour 24
Population: Biomarker population-all treated participants who had any available biomarker data
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 | Arm 4: Heathy Participants
Number analyzed (Participants) | 15 | 15 | 15 | 11
Percent Change
  On-treatment Day 1, Hour 2, Low Shear | 10.0 (260.3) | 538.6 (1803.3) | 104.2 (383.5) | -14.9 (50.2)
  On-treatment Day 1, Hour 2, High Shear | -23.0 (24.1) | -18.4 (27.5) | -24.2 (17.2) | -27.7 (24.4)
  Post-treatment Day 2, Hour 24, Low Shear: number analyzed (Participants) | 15 | 15 | 15 | 10
  Post-treatment Day 2, Hour 24, Low Shear | 20.7 (134.6) | 579.6 (2125.4) | 31.0 (130.0) | -2.5 (41.6)
  Post-treatment Day 2, Hour 24, High Shear: number analyzed (Participants) | 15 | 15 | 15 | 10
  Post-treatment Day 2, Hour 24, High Shear | -4.8 (30.0) | -3.5 (67.1) | -10.6 (24.0) | -23.0 (22.2)

2. Secondary Outcome: Number of Participants Experiencing Abnormal Vital Signs
Description: The number of participants with abnormal vital sign values. The criteria used for classifying vital sign results as markedly abnormal is listed below. Baseline is defined as the last non-missing result with a collection date-time less than the date-time of the first dose of study medication. For Treatment Arms 1, 2, and 3, a baseline chamber run was performed approximately 2 hours after background therapy (ticagrelor, aspirin, or ticagrelor + aspirin) and prior to BMS-986141 administration. A second chamber run was performed 2 hours following oral administration of BMS-986141. For Treatment Arm 4, a baseline chamber run was performed prior to BMS-986141 administration. A second chamber run was performed 2 hours following oral administration of BMS-986141. Participants received background therapy before the final chamber run, and the final chamber run was performed on Day 2, approximately 24 hours after BMS-986141 dosing.
Time Frame: Vital signs will be collected at check-in and prior to and after each chamber assessment on Days 1 and 2
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Arm 4: Heathy Participants: Heathy Participants
Arm/Group | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 | Arm 4: Heathy Participants
Number analyzed (Participants) | 16 | 15 | 16 | 11
Participants
  DIASTOLIC BLOOD PRESSURE (MMHG) Day 1 > 90 AND CHANGE FROM BASELINE > 10: number analyzed (Participants) | 16 | 14 | 15 | 11
  DIASTOLIC BLOOD PRESSURE (MMHG) Day 1 > 90 AND CHANGE FROM BASELINE > 10 | 2 | 0 | 0 | 0
  DIASTOLIC BLOOD PRESSURE (MMHG) Pre-Chamber Run > 90 AND CHANGE FROM BASELINE > 10: number analyzed (Participants) | 16 | 15 | 15 | 11
  DIASTOLIC BLOOD PRESSURE (MMHG) Pre-Chamber Run > 90 AND CHANGE FROM BASELINE > 10 | 2 | 0 | 0 | 0
  DIASTOLIC BLOOD PRESSURE (MMHG) Post-Chamber Run < 55 AND CHANGE FROM BASELINE < -10: number analyzed (Participants) | 15 | 15 | 15 | 11
  DIASTOLIC BLOOD PRESSURE (MMHG) Post-Chamber Run < 55 AND CHANGE FROM BASELINE < -10 | 0 | 0 | 1 | 0
  DIASTOLIC BLOOD PRESSURE (MMHG) Post-Chamber Run > 90 AND CHANGE FROM BASELINE > 10: number analyzed (Participants) | 15 | 15 | 15 | 11
  DIASTOLIC BLOOD PRESSURE (MMHG) Post-Chamber Run > 90 AND CHANGE FROM BASELINE > 10 | 1 | 0 | 0 | 0
  DIASTOLIC BLOOD PRESSURE (MMHG) 2 hours Pre-Chamber Run > 90 AND CHANGE FROM BASELINE > 10: number analyzed (Participants) | 15 | 15 | 15 | 11
  DIASTOLIC BLOOD PRESSURE (MMHG) 2 hours Pre-Chamber Run > 90 AND CHANGE FROM BASELINE > 10 | 1 | 0 | 0 | 0
  DIASTOLIC BLOOD PRESSURE (MMHG) 2 hours Post-Chamber Run > 90 AND CHANGE FROM BASELINE > 10: number analyzed (Participants) | 15 | 14 | 15 | 11
  DIASTOLIC BLOOD PRESSURE (MMHG) 2 hours Post-Chamber Run > 90 AND CHANGE FROM BASELINE > 10 | 0 | 0 | 1 | 1
  DIASTOLIC BLOOD PRESSURE (MMHG) 24 hours Pre-Chamber Run > 90 AND CHANGE FROM BASELINE > 10: number analyzed (Participants) | 15 | 15 | 15 | 11
  DIASTOLIC BLOOD PRESSURE (MMHG) 24 hours Pre-Chamber Run > 90 AND CHANGE FROM BASELINE > 10 | 2 | 1 | 0 | 0
  DIASTOLIC BLOOD PRESSURE (MMHG) 24 hours Pre-Chamber Run < 55 AND CHANGE FROM BASELINE < -10: number analyzed (Participants) | 15 | 15 | 15 | 11
  DIASTOLIC BLOOD PRESSURE (MMHG) 24 hours Pre-Chamber Run < 55 AND CHANGE FROM BASELINE < -10 | 0 | 1 | 0 | 0
  HEART RATE (BEATS/MIN) Day 1 HR < 55 AND CHANGE FROM BASELINE < -15: number analyzed (Participants) | 16 | 14 | 15 | 11
  HEART RATE (BEATS/MIN) Day 1 HR < 55 AND CHANGE FROM BASELINE < -15 | 0 | 1 | 0 | 0
  HEART RATE (BEATS/MIN) Pre-Chamber Run HR < 55 AND CHANGE FROM BASELINE < -15: number analyzed (Participants) | 16 | 15 | 15 | 11
  HEART RATE (BEATS/MIN) Pre-Chamber Run HR < 55 AND CHANGE FROM BASELINE < -15 | 0 | 1 | 0 | 0
  HEART RATE (BEATS/MIN) Post-Chamber Run HR < 55 AND CHANGE FROM BASELINE < -15: number analyzed (Participants) | 15 | 15 | 15 | 11
  HEART RATE (BEATS/MIN) Post-Chamber Run HR < 55 AND CHANGE FROM BASELINE < -15 | 0 | 1 | 0 | 0
  HEART RATE (BEATS/MIN) 2 Hour Pre-Chamber Run HR < 55 AND CHANGE FROM BASELINE < -15: number analyzed (Participants) | 15 | 15 | 15 | 11
  HEART RATE (BEATS/MIN) 2 Hour Pre-Chamber Run HR < 55 AND CHANGE FROM BASELINE < -15 | 0 | 1 | 0 | 0
  HEART RATE (BEATS/MIN) 2 Hour Post-Chamber Run HR < 55 AND CHANGE FROM BASELINE < -15: number analyzed (Participants) | 15 | 14 | 15 | 11
  HEART RATE (BEATS/MIN) 2 Hour Post-Chamber Run HR < 55 AND CHANGE FROM BASELINE < -15 | 0 | 1 | 0 | 0
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 Day 1: number analyzed (Participants) | 16 | 14 | 15 | 11
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 Day 1 | 1 | 0 | 3 | 0
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 Pre-Chamber Run: number analyzed (Participants) | 16 | 15 | 15 | 11
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 Pre-Chamber Run | 4 | 0 | 3 | 0
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 Post-Chamber Run: number analyzed (Participants) | 15 | 15 | 15 | 11
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 Post-Chamber Run | 5 | 3 | 4 | 0
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 2 Hour Pre-Chamber Run: number analyzed (Participants) | 15 | 15 | 15 | 11
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 2 Hour Pre-Chamber Run | 2 | 4 | 4 | 1
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 2 Hour Post-Chamber Run: number analyzed (Participants) | 15 | 14 | 15 | 11
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 2 Hour Post-Chamber Run | 2 | 2 | 2 | 0
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 24 Hour Pre-Chamber Run: number analyzed (Participants) | 15 | 15 | 15 | 11
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 24 Hour Pre-Chamber Run | 1 | 3 | 6 | 0
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 24 Hour Post-Chamber Run: number analyzed (Participants) | 15 | 15 | 15 | 11
  RESPIRATORY RATE (BREATHS/MIN) > 16 OR CHANGE FROM BASELINE > 10 24 Hour Post-Chamber Run | 0 | 2 | 8 | 1
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 Day 1 Pre-Chamber Run: number analyzed (Participants) | 16 | 15 | 15 | 11
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 Day 1 Pre-Chamber Run | 1 | 0 | 1 | 0
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 2 Hour Pre-Chamber Run: number analyzed (Participants) | 15 | 15 | 15 | 11
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 2 Hour Pre-Chamber Run | 1 | 0 | 1 | 0
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 2 Hour Post-Chamber Run: number analyzed (Participants) | 15 | 14 | 15 | 11
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 2 Hour Post-Chamber Run | 2 | 0 | 0 | 0
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 24 Hour Pre-Chamber Run: number analyzed (Participants) | 15 | 15 | 15 | 11
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 24 Hour Pre-Chamber Run | 0 | 1 | 0 | 0
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 24 Hour Post-Chamber Run: number analyzed (Participants) | 15 | 15 | 15 | 11
  SYSTOLIC BLOOD PRESSURE (MMHG) > 140 AND CHANGE FROM BASELINE > 20 24 Hour Post-Chamber Run | 0 | 1 | 0 | 0
  TEMPERATURE (C) > 38.3 OR CHANGE FROM BASELINE > 1.6 Day 1: number analyzed (Participants) | 16 | 14 | 15 | 11
  TEMPERATURE (C) > 38.3 OR CHANGE FROM BASELINE > 1.6 Day 1 | 1 | 0 | 0 | 0
  TEMPERATURE (C) > 38.3 OR CHANGE FROM BASELINE > 1.6 Pre-Chamber Run: number analyzed (Participants) | 16 | 15 | 15 | 11
  TEMPERATURE (C) > 38.3 OR CHANGE FROM BASELINE > 1.6 Pre-Chamber Run | 1 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Experiencing Abnormal Electrocardiogram (ECG) Values
Description: The number of participants with abnormal electrocardiogram values. The criteria used for classifying electrocardiogram results as markedly abnormal is listed below. The 2-hour and 24-hour ECGs should are performed prior to the Badimon Chamber run. Baseline is defined as the last non-missing result with a collection date-time less than the date-time of the first dose of study medication.
Time Frame: Electrocardiograms were collected at check-in, and 2 and 24 hours after dosing
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 | Arm 4: Heathy Participants
Number analyzed (Participants) | 16 | 15 | 16 | 11
Participants
  PR INTERVAL, AGGREGATE (MSEC) Baseline <210 | 5 | 6 | 1 | 0
  PR INTERVAL, AGGREGATE (MSEC) Baseline >=210 | 0 | 0 | 0 | 0
  PR INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 <210: number analyzed (Participants) | 15 | 15 | 15 | 11
  PR INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 <210 | 4 | 5 | 1 | 0
  PR INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 >=210: number analyzed (Participants) | 15 | 15 | 15 | 11
  PR INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 >=210 | 1 | 1 | 0 | 0
  QRS DURATION, AGGREGATE (MSEC) Baseline <120 | 5 | 6 | 1 | 0
  QRS DURATION, AGGREGATE (MSEC) Baseline >=120 | 0 | 0 | 0 | 0
  QRS DURATION, AGGREGATE (MSEC) Day 2, Hour 24 <120: number analyzed (Participants) | 15 | 15 | 15 | 11
  QRS DURATION, AGGREGATE (MSEC) Day 2, Hour 24 <120 | 5 | 6 | 1 | 0
  QRS DURATION, AGGREGATE (MSEC) Day 2, Hour 24 >=120: number analyzed (Participants) | 15 | 15 | 15 | 11
  QRS DURATION, AGGREGATE (MSEC) Day 2, Hour 24 >=120 | 0 | 0 | 0 | 0
  QT INTERVAL, AGGREGATE (MSEC) Baseline <500 | 5 | 6 | 1 | 0
  QT INTERVAL, AGGREGATE (MSEC) Baseline >=500 | 0 | 0 | 0 | 0
  QT INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 <500: number analyzed (Participants) | 15 | 15 | 15 | 11
  QT INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 <500 | 5 | 6 | 1 | 0
  QT INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 >=500: number analyzed (Participants) | 15 | 15 | 15 | 11
  QT INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 >=500 | 0 | 0 | 0 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) Baseline <450 | 5 | 6 | 1 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) Baseline >=450 | 0 | 0 | 0 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 <450: number analyzed (Participants) | 15 | 15 | 15 | 11
  QTCF INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 <450 | 5 | 5 | 1 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 >=450: number analyzed (Participants) | 15 | 15 | 15 | 11
  QTCF INTERVAL, AGGREGATE (MSEC) Day 2, Hour 24 >=450 | 0 | 1 | 0 | 0

4. Secondary Outcome: Number of Participants Experiencing Clinical Lab Abnormalities
Description: The number of participants with abnormal clinical laboratory results. The criteria used for classifying laboratory test results as markedly abnormal is listed below.
Time Frame: From baseline up to 24 hours post dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 | Arm 4: Heathy Participants
Number analyzed (Participants) | 16 | 15 | 16 | 11
Participants
  HEMOGLOBIN (G/DL)-Abnormal Low | 0 | 2 | 0 | 0
  HEMATOCRIT (%)-Abnormal Low | 0 | 2 | 0 | 0
  ERYTHROCYTES (X10*6 C/UL)-Abnormal Low | 0 | 1 | 0 | 1
  LEUKOCYTES (X10*3 C/UL)-Abnormal Low | 0 | 0 | 1 | 1
  LEUKOCYTES (X10*3 C/UL)-Abnormal High | 0 | 1 | 0 | 0
  NEUTROPHILS (ABSOLUTE) (X10*3 C/UL)-Abnormal Low | 0 | 0 | 0 | 1
  BLOOD UREA NITROGEN (MG/DL)-Abnormal High | 3 | 3 | 0 | 0
  POTASSIUM, SERUM (MEQ/L)-Abnormal Low | 0 | 1 | 0 | 0
  CHLORIDE, SERUM (MEQ/L)-Abnormal High | 0 | 1 | 0 | 0
  CALCIUM, TOTAL (MG/DL)-Abnormal Low | 0 | 1 | 0 | 1
  PHOSPHORUS, INORGANIC (MG/DL)-Abnormal Low | 0 | 1 | 0 | 0
  MAGNESIUM, SERUM (MEQ/L)-Abnormal Low | 0 | 1 | 0 | 0
  GLUCOSE, FASTING SERUM (MG/DL)-Abnormal Low | 0 | 0 | 1 | 0
  GLUCOSE, FASTING SERUM (MG/DL)-Abnormal High | 2 | 0 | 1 | 0
  PROTEIN, TOTAL (G/DL) -Abnormal Low | 0 | 1 | 0 | 1
  ALBUMIN (G/DL)-Abnormal Low | 1 | 2 | 1 | 1
  CREATINE KINASE (U/L)-Abnormal High | 1 | 1 | 0 | 0
  PROTEIN, URINE (N/A)-Abnormal High | 1 | 0 | 0 | 0
  GLUCOSE, URINE (N/A)-Abnormal High | 1 | 0 | 0 | 0
  BLOOD, URINE (N/A)-Abnormal High | 1 | 1 | 1 | 0
  RBC, URINE (HPF)-Abnormal High | 0 | 0 | 2 | 0
  WBC, URINE (HPF)-Abnormal High | 1 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 8 days post last dose
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 | Arm 4: Heathy Participants
Number analyzed (Participants) | 16 | 15 | 16 | 11
Participants | 6 | 0 | 4 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from first dose to 30 days following last dose, up to approximately 32 days.
Arm/Group | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 | Arm 4: Heathy Participants
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 6/16 | 0/15 | 4/16 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: 90 mg Ticagrelor + 4 mg BMS-986141 (N=16) | Arm 2: 75 mg Aspirin + 4 mg BMS-986141 (N=15) | Arm 3: 90 mg Ticagrelor + 75 mg Aspirin + 4 mg BMS-986141 (N=16) | Arm 4: Heathy Participants (N=11)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT05093790/Prot_SAP_000.pdf